CLINICAL TRIAL: NCT02833857
Title: An Open-label, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Etelcalcetide (AMG 416) in Paediatric Subjects Aged 2 to Less Than 18 Years With Secondary Hyperparathyroidism (sHPT) Receiving Maintenance Haemodialysis
Brief Title: A Single-dose Study in Paediatric Patients Aged 2 to Less Than 18 Years With Secondary Hyperparathyroidism (sHPT) Receiving Haemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140336; 2015-005051-28 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-07-14 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease, Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism, chronic kidney disease, hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etelcalcetide (Experimental): Participants received a single, intravenous (IV) bolus administration of 0.035 mg/kg etelcalcetide at the end of hemodialysis on study day 1.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — A single IV-bolus dose of 0.035 mg/kg etelcalcetide into the venous line of the dialysis circuit at the end of a hemodialysis session.
  Other Names: AMG 416; Parsabiv

SUMMARY:
This is a study to evaluate the safety and pharmacokinetics in pediatric patients with secondary hyperparathyroidism receiving a single dose of etelcalcetide at the end of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent has provided informed consent and subject has provided assent
* Children Age 2 to less than 18 years
* Diagnosed with chronic kidney disease
* Diagnosed with secondary hyperparathyroidism receiving hemodialysis,
* Weighing at least 7 kg
* Laboratory results within specified range.

Exclusion Criteria:

* Currently receiving treatment in another investigation device or drug study
* Subject has received cinacalcet therapy within 30 days
* History of prolongation QT interval
* Subject is taking any medications that are on the QT prolongation medication list
* Electrocardiograph (ECG) measurements within specified range.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Louisville, Kentucky
  - Research Site, Kansas City, Missouri
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Germany (4):
  - Research Site, Cologne
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Marburg
- Research Site, Vilinus, Lithuania
- Research Site, Krakow, Poland
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Sohn W, Salusky IB, Schmitt CP, Taylan C, Walle JV, Ngang J, Yan L, Kroenke M, Warady BA. Phase 1, single-dose study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of etelcalcetide in pediatric patients with secondary hyperparathyroidism receiving hemodialysis. Pediatr Nephrol. 2021 Jan;36(1):133-142. doi: 10.1007/s00467-020-04599-z. Epub 2020 Jul 9. PMID 32647975
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 centers in the United States, United Kingdom, and the European Union. Participants were enrolled from 14 March 2017 to 01 October 2018.
Period: Overall Study
Arm/Group | Etelcalcetide
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (4.3)
Age, Customized [Count of Participants; unit: Participants]
  Children (2 to 11 years) | 5
  Adolescents (12 to 17 years) | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black (or African American) | 2
  White | 9
Serum Corrected Calcium Concentration [Mean (Standard Deviation); unit: mmol/L] — When albumin was less than 4.0 mg/dL, the calcium concentration was corrected according to the formula: cCa (mmol/L) = measured total serum calcium (mmol/L) + 0.02 (40 - serum albumin [g/L]).
  mmol/L | 2.42 (0.08)
Serum Phosphorus Concentration [Mean (Standard Deviation); unit: mmol/L] — Population: Participants with available data
  mmol/L
    number analyzed (Participants) | 10
    (all) | 1.79 (0.45)
Serum Potassium Concentration [Mean (Standard Deviation); unit: mmol/L] | 4.77 (0.55)
Serum Intact Parathyroid Hormone Concentration [Mean (Standard Deviation); unit: pmol/L] | 66.10 (57.57)
Serum Calcium Concentration [Mean (Standard Deviation); unit: mmol/L] | 2.41 (0.08)
Serum Ionized Calcium Concentration [Mean (Standard Deviation); unit: mmol/L] | 1.16 (0.07)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 87.4 (9.9)
Temperature [Mean (Standard Deviation); unit: degrees celsius] | 36.6 (0.3)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic blood pressure | 119.4 (15.9)
  Diastolic blood pressure | 66.7 (15.1)
PR Interval [Mean (Standard Deviation); unit: ms] — The PR interval is measured using electrocardiography (ECG) and is the period from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex (the onset of ventricular depolarization); it is normally between 120 and 200 milliseconds (ms) in duration.
  ms | 133.8 (8.7)
QRS Interval [Mean (Standard Deviation); unit: ms] — The QRS interval measured during ECG, denotes depolarization of the ventricles, between the beginning of the Q wave and the end of the S wave.
  ms | 82.0 (10.9)
QT Interval [Mean (Standard Deviation); unit: ms] — The QT interval measured during ECG is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QT interval represents electrical depolarization and repolarization of the ventricles.
  ms | 363.5 (26.2)
Corrected (Bazett) QT Interval (QTcB) [Mean (Standard Deviation); unit: ms] | 424.2 (29.1)
Corrected (Fridericia) QT Interval (QTcF) [Mean (Standard Deviation); unit: ms] | 402.7 (26.1)

OUTCOME MEASURES:

1. Primary Outcome: Common Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event is any adverse event (AE) that begins or worsens after the initial dose of study drug (etelcalcetide) and up to 30 days after the last dose.
  Common adverse events were defined as adverse events occurring in at least 2 participants.
  The Medical Dictionary for Regulatory Activities (MedDRA) version 21.0 was used for coding all adverse events.
Time Frame: 30 days
Population: Participants who received at least 1 dose of etelcalcetide (safety analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
Participants
  Headache | 2
  Calcium ionised decreased | 2
  Hypotension | 2

2. Primary Outcome: Change From Baseline in Serum Corrected Calcium Concentration Over Time
Description: When albumin was less than 4.0 mg/dL, the calcium concentration was corrected according to the formula: cCa (mmol/L) = measured total serum calcium (mmol/L) + 0.02 (40 - serum albumin [g/L]).
Time Frame: Baseline and Day 1, 4 hours postdose, day 3, day 8, day 10, and day 30 (end of study)
Population: Treated participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmol/L
  Day 1, 4 hours: number analyzed (Participants) | 10
  Day 1, 4 hours | -0.03 (0.12)
  Day 3 | -0.03 (0.08)
  Day 8 | 0.03 (0.09)
  Day 10 | 0.03 (0.07)
  Day 30 | -0.01 (0.16)

3. Primary Outcome: Change From Baseline in Serum Phosphorus Concentration at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmol/L | 0.08 (0.31)

4. Primary Outcome: Change From Baseline in Serum Potassium Concentration at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmol/L | 0.45 (1.21)

5. Primary Outcome: Change From Baseline in Intact Parathyroid Hormone (iPTH) Levels Over Time
Time Frame: Baseline and day 1, 4 hours postdose, day 3, day 8, day 10, and day 30 (end of study)
Population: Treated participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
pmol/L
  Day 1, 4 hours: number analyzed (Participants) | 10
  Day 1, 4 hours | -29.44 (37.16)
  Day 3 | -14.81 (37.81)
  Day 8 | -10.20 (38.16)
  Day 10 | -4.68 (37.92)
  Day 30 | -19.81 (51.29)

6. Primary Outcome: Change From Baseline in Heart Rate at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
beats/minute | -4.5 (9.3)

7. Primary Outcome: Change From Baseline in Temperature at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
degrees celsius | 0.1 (0.4)

8. Primary Outcome: Change From Baseline in Blood Pressure at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmHg
  Systolic blood pressure | 0.2 (17.5)
  Diastolic blood pressure | 3.8 (8.5)

9. Primary Outcome: Change From Baseline in PR Interval at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ms | -3.6 (13.9)

10. Primary Outcome: Change From Baseline in QRS Interval at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ms | -2.6 (6.8)

11. Primary Outcome: Change From Baseline in QT Interval at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ms | 2.8 (21.6)

12. Primary Outcome: Change From Baseline in Corrected (Bazett) QT Interval at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ms | -2.1 (32.2)

13. Primary Outcome: Change From Baseline in Corrected (Fridericia) QT Interval at End of Study
Time Frame: Baseline and day 30 (end of study)
Population: Treated participants
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ms | -0.5 (23.3)

14. Secondary Outcome: Change From Baseline in Serum Total Calcium Concentration
Time Frame: Baseline and Day 1, 4 hours postdose, day 3, day 8, day 10, and day 30 (end of study)
Population: Treated participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmol/L
  Day 1, 4 hours: number analyzed (Participants) | 10
  Day 1, 4 hours | -0.02 (0.12)
  Day 3 | -0.02 (0.08)
  Day 8 | 0.03 (0.08)
  Day 10 | 0.02 (0.08)
  Day 30 | -0.01 (0.16)

15. Secondary Outcome: Change From Baseline in Serum Ionized Calcium Concentration
Time Frame: Baseline and Day 1, 4 hours postdose, day 3, day 8, day 10, and day 30 (end of study)
Population: Treated participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
mmol/L
  Day 1, 4 hours: number analyzed (Participants) | 10
  Day 1, 4 hours | -0.05 (0.13)
  Day 3: number analyzed (Participants) | 10
  Day 3 | -0.01 (0.08)
  Day 8 | 0.02 (0.07)
  Day 10 | 0.01 (0.06)
  Day 30 | 0.03 (0.06)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Etelcalcetide
Description: Plasma etelcalcetide concentrations were measured using a validated high performance liquid chromatography assay. The lower limit of quantitation was 0.200 ng/mL.
Time Frame: 10 minutes, 4 hours, and 3, 5, 8, 10, and 30 days postdose
Population: The pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
ng/mL | 50.8 (29.3)

17. Secondary Outcome: Time to Maximum Concentration (Tmax) of Etelcalcetide
Description: as for outcome 16
Time Frame: 10 minutes, 4 hours, and 3, 5, 8, 10, and 30 days postdose
Population: The pharmacokinetic concentration analysis set was composed of all participants who received etelcalcetide and had at least 1 pharmacokinetic sample collected.
Measure: Median (Full Range); unit: hours
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
hours | 0.17 [0.17 to 0.33]

18. Secondary Outcome: Area Under the Plasma Etelcalcetide Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: Plasma etelcalcetide concentrations were measured using a validated high performance liquid chromatography assay. The lower limit of quantitation was 0.200 ng/mL.
  Area under the curve for plasma etelcalcetide from time zero to the last quantifiable concentration (AUClast) was estimated using the linear trapezoidal method.
Time Frame: 10 minutes, 4 hours, and 3, 5, 8, 10, and 30 days postdose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
hr*ng/mL | 1360 (1110)

19. Secondary Outcome: Area Under the Plasma Etelcalcetide Concentration-Time Curve From Time Zero Infinity (AUCinf)
Description: Plasma etelcalcetide concentrations were measured using a validated high performance liquid chromatography assay. The lower limit of quantitation was 0.200 ng/mL.
  Area under the concentration-time curve from time zero to infinite time (AUCinf) was estimated using the linear trapezoidal method.
Time Frame: 10 minutes, 4 hours, and 3, 5, 8, 10, and 30 days postdose
Population: Pharmacokinetic analysis set with available AUCinf data
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 7
hr*ng/mL | 1700 (1420)

20. Secondary Outcome: Terminal Half-life (T1/2,z) of Etelcalcetide
Description: Plasma etelcalcetide concentrations were measured using a validated high performance liquid chromatography assay. The lower limit of quantitation was 0.200 ng/mL.
  Terminal half life of plasma etelcalcetide (t1/2,z) was calculated as t1/2,z = ln(2)/λz, where λz is the first-order terminal rate constant estimated by linear regression of the terminal log-linear phase.
Time Frame: 10 minutes, 4 hours, and 3, 5, 8, 10, and 30 days postdose
Population: Pharmacokinetic analysis set with available T1/2,z data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 7
days | 5.77 (2.66)

21. Secondary Outcome: Number of Participants Who Developed Anti-etelcalcetide Binding Antibodies
Description: Samples were collected predose and at end of study (day 30) and tested for anti etelcalcetide binding antibodies using a validated immunoassay.
  Developing antibody binding was defined as participants who were binding antibody positive postbaseline with a negative result at baseline.
Time Frame: Baseline and day 30
Population: Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
Participants | 2

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event is any adverse event that begins or worsens after the initial dose of study drug (etelcalcetide) and up to 30 days after the last dose. The severity of each adverse event was graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, where Grade 1 = Mild (asymptomatic or mild symptoms), Grade 2 = Moderate (minimal, local or noninvasive intervention indicated), Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated, Grade 4 = Life-threatening consequences; urgent intervention indicated, and Grade 5 = Death related to AE.
Time Frame: 30 days
Population: All Treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 11
Participants
  Any adverse event | 6
  Adverse events ≥ grade 3 | 2
  Adverse events ≥ grade 4 | 0
  Serious adverse events | 0
  AEs leading to discontinuation of etelcalcetide | 0
  Fatal adverse events | 0
  Treatment-related adverse events | 0
  Treatment-related AEs ≥ grade 3 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Etelcalcetide: Participants received a single, intravenous bolus administration of 0.035 mg/kg etelcalcetide at the end of hemodialysis on study day 1.
Arm/Group | Etelcalcetide
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=11)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Calcium ionised decreased (Investigations) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Gastrostomy (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02833857/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02833857/SAP_001.pdf